CLINICAL TRIAL: NCT06043661
Title: An Evaluation of a Circulating Tumor Cell-based Test (TriNetra™-Breast) for Breast Cancer Screening in Women Aged 40 and Above
Brief Title: Early Detection of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Datar Cancer Genetics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HUM00217725
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms
Keywords: Early Detection; Mammography; Circulating Tumor Cells; Cancer Screening
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BI-RADS score 1 or 2 or 3 (Cohort A): Subjects with a standard risk of breast cancer aged 40 years and above at the time of mammography with the BI-RADS score 1 or 2 or 3
- BI-RADS score 4 or 5 (Cohort B): Subjects aged 40 years and above at the time of mammography with the BI-RADS score 4 or 5

SUMMARY:
The TriNetra™ Breast test is intended for use as a breast cancer screening test that evaluates Circulating Tumor Cells (CTCs) associated with breast cancer. The TriNetra™Breast test should be a useful breast cancer screening option for asymptomatic women 40 years of age and older.

This pivotal study is designed to provide evidence of test performance and to demonstrate its safety in the intended use population in the USA.

DETAILED DESCRIPTION:
This prospective, case-cohort study evaluates the sensitivity and specificity of the TriNetra™-Breast test for breast cancer (adenocarcinoma) screening in women aged 40 years and older. Approximately 700 subjects will be enrolled in one of the two non-overlapping cohorts in this study. Cohort A will enroll about 500 subjects with a standard risk of breast cancer who fulfill the enrollment criteria. Cohort B will enroll approximately 200 subjects with a mammogram result of BI-RADS 4 or 5.

The results of TriNetra™ -Breast will be compared with the results of mammography. The corresponding diagnostic biopsy pathology results obtained as the standard of care will be correlated with test results to confirm the performance estimates (when indicated). Mammography will be the reference standard of evaluation of breast screening status for cohort A. Histopathology report will be the reference standard to evaluate the malignant or non-malignant clinical status for cohort B. Availability of histopathological results is mandatory for the evaluation of cohort B.

ELIGIBILITY:
Inclusion Criteria:

A). For Cohort A (500 subjects are targeted to enroll)

1. No prior diagnosis of (any) cancer
2. Women aged 40 years and above at the time of mammography
3. Provision of signed informed consent
4. Capable of providing adequate health history
5. No co-morbidity which could impair study participation or sample collection
6. Blood draw within sixty (60) days of performance of screening mammography
7. A redacted/deidentified mammography report will be available and provided
8. If any prior mammography was performed, the BI-RADS score should be 1 or 2 or 3
9. Willingness to accept follow-up contact every 6 months for up to 2 years.
10. Agreeable to share any future biopsy or imaging data for a maximum of 2 years from study blood draw.

B). For Cohort B (BI-RADS 4 and 5) (200 subjects are targeted to enroll)

1. No prior diagnosis of (any) cancer
2. Women aged 40 years and above at the time of mammography
3. Provision of signed informed consent
4. Current mammography indicating BI-RADS 4a,4b, 4c, or 5
5. Capable of providing adequate health history
6. No co-morbidity which could impair study participation or sample collection
7. Blood draw within sixty (60) days of mammography and prior to biopsy of the breast
8. Yet to undergo tissue diagnostic procedure for breast lesion such as fine needle, core, or excisional biopsy
9. A redacted/deidentified mammography report and redacted/de-identified pathology report will be available and provided
10. Willingness to accept follow-up contact every 6 months for up to 2 years.
11. Agreeable to share any future repeat biopsy or imaging data for a maximum of 2 years from study blood draw.

C). Exclusion Criteria

1. Prior diagnosis of (any) cancer
2. Subjects who are receiving any investigational agent.
3. Pregnant women are excluded from this study
4. Breastfeeding women are excluded from this study
5. Blood transfusion within 30 days prior to screening,
6. Subject has any condition that in the opinion of the investigator should preclude participation in the study.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of women aged 40 years and older. The target enrollment will be approximately 700 subjects, who will be divided into two non-overlapping cohorts.
  All subjects enrolled in the study will undergo a blood draw for TriNetraTM Breast around the time of mammography. The blood draw will have to be performed no more than 60 days after the mammography and before the breast biopsy (Cohort B).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the sensitivity and specificity of TriNetra Breast for breast cancer screening in women 40 years and older, using mammography and histopathology confirmed diagnosis (when relevant) as the reference methods. | 2 years
  The study evaluates the clinical sensitivity and specificity of the TriNetra Breast in Mammography-Negative (BIRAD 1/2/3) and Mammography-Positive (BIRAD 4/5) Cohorts

SECONDARY OUTCOMES:
The Positive Predictive Values (PPV) and Negative Predictive Values (NPV) | 2 years
  The study evaluates the PPV and NPV of the TriNetra Breast for breast cancer screening in women 40 years and older, using mammography and histopathology confirmed diagnosis (when relevant) as the reference methods.
Detection rates by TNM stage | 2 years
  The study evaluates the detection rates (sensitivity in %) by TNM stage for the TriNetra Breast test, using surgical pathology evaluation as a reference.
Clinical performance in dense breast findings on mammography | 2 years
  The study evaluates the clinical sensitivity and specificity (in %) for the TriNetra Breast test in dense breast findings on mammography
Sensitivity and specificity for ductal carcinoma in situ (DCIS) detection | 2 years
  The study evaluates the clinical sensitivity and specificity (in %) for the TriNetra Breast test in ductal carcinoma in situ (DCIS) detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Rogel Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Crook T, Leonard R, Mokbel K, Thompson A, Michell M, Page R, Vaid A, Mehrotra R, Ranade A, Limaye S, Patil D, Akolkar D, Datta V, Fulmali P, Apurwa S, Schuster S, Srinivasan A, Datar R. Accurate Screening for Early-Stage Breast Cancer by Detection and Profiling of Circulating Tumor Cells. Cancers (Basel). 2022 Jul 9;14(14):3341. doi: 10.3390/cancers14143341. PMID 35884402